CLINICAL TRIAL: NCT02501811
Title: A Phase II, Randomized, Placebo-Controlled Study of the Safety, Feasibility, & Efficacy of Autologous Mesenchymal Stem Cells & C-kit+ Cardiac Stem Cells, Alone or in Combination, Administered Transendocardially in Subjects With Ischemic HF
Brief Title: Combination of Mesenchymal and C-kit+ Cardiac Stem Cells as Regenerative Therapy for Heart Failure
Acronym: CONCERT-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barry R Davis, Professor of Biostatistics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-SPH-15-0413; 5UM1HL087318 (NIH)
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Heart Failure; Ischemia; Autologous Stem Cells; LV dysfunction; Mesenchymal Stem Cells; c-kit+ Cells; Combination Cell Therapy; LV function; Functional status
MeSH Terms: conditions — Heart Failure; Ischemia; Ventricular Dysfunction, Left | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mesenchymal Stem Cells (MSC) (Experimental): Target dose of 150 million MSCs
  Interventions: Biological: Mesenchymal Stem Cells (MSC)
- c-kit+ cells (Experimental): Target dose of 5 million c-kit+ cells
  Interventions: Biological: c-kit+ cells
- Combination Cells (MSC and c-kit+ cells) (Experimental): Target dose of 150 million MSCs and 5 million c-kit+ cells
  Interventions: Biological: Mesenchymal Stem Cells (MSC); Biological: c-kit+ cells
- Placebo (Plasmalyte A) (Placebo Comparator): Plasmalyte A
  Interventions: Biological: Placebo (Plasmalyte A)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSC) — 15 transendocardial injections of 0.4ml MSCs administered to the left ventricle via NOGA Myostar injection catheter (single procedure)
  Arms: Combination Cells (MSC and c-kit+ cells); Mesenchymal Stem Cells (MSC)
Biological: c-kit+ cells — 15 transendocardial injections of 0.4ml c-kit+ cells administered to the left ventricle via NOGA Myostar injection catheter (single procedure)
  Arms: Combination Cells (MSC and c-kit+ cells); c-kit+ cells
Biological: Placebo (Plasmalyte A) — 15 transendocardial injections of 0.4ml placebo administered to the left ventricle via NOGA Myostar injection catheter (single procedure)
  Other Names: Plasmalyte A
  Arms: Placebo (Plasmalyte A)

SUMMARY:
This is a phase II, randomized, placebo-controlled clinical trial designed to assess feasibility, safety, and effect of autologous bone marrow-derived mesenchymal stem cells (MSCs) and c-kit+ cells both alone and in combination (Combo), compared to placebo (cell-free Plasmalyte-A medium) as well as each other, administered by transendocardial injection in subjects with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled clinical trial designed to evaluate the feasibility, safety, and effect of Combo, MSCs alone, and c-kit+ cells alone compared with placebo as well as each other in subjects with heart failure of ischemic etiology. Following a successful lead-in phase, a total of one hundred forty-four (144) subjects will be randomized (1:1:1:1) to receive Combo, MSCs, c-kit+ cells, or placebo. After randomization, baseline imaging, relevant harvest procedures, and study product injection, subjects will be followed up at 1 day, 1 week, 1 month, 3 months, 6 months and 12 months post study product injection. All subjects will receive study product injection (cells or placebo) using the NOGA® XP Mapping and Navigation System. Subjects will have delayed-enhanced magnetic resonance imaging (DEMRI) scans to assess scar size and LV function and structure at baseline and at 6 and 12 months post study product administration. All endpoints will be assessed at the 6 and 12 month visits which will occur 180 ±30 days and 365 ±30 days respectively from the day of study product injection (Day 0). For the purpose of the endpoint analysis and safety evaluations, the Investigators will utilize an "intention-to-treat" study population, however an as treated analysis will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 21 and <80 years of age
2. Have documented coronary artery disease (CAD) with evidence of myocardial injury, LV dysfunction, and clinical evidence of HF
3. Have a "detectable" area of myocardial injury defined as ≥ 5% LV involvement (infarct volume) and any subendocardial involvement by cMRI
4. Have an EF ≤ 40% by cMRI
5. Be receiving guideline-driven medical therapy for heart failure at stable and tolerated doses for ≥ 1 month prior to consent. For beta-blockade "stable" is defined as no greater than a 50% reduction in dose or no more than a 100% increase in dose.
6. Be a candidate for cardiac catheterization
7. Have NYHA class I, II, or III heart failure symptoms
8. If a female of childbearing potential, be willing to use one form of birth control for the duration of the study, and undergo a pregnancy test at baseline and within 36 hours prior to injection

Exclusion Criteria:

1. Indication for standard-of-care surgery (including valve surgery, placement of left-ventricular assist device, or imminent heart transplantation), coronary artery bypass grafting (CABG) procedure, and/or percutaneous coronary intervention (PCI) for the treatment of ischemic and/or valvular heart disease. Subjects who require or undergo PCI should undergo these procedures a minimum of 3 months in advance of randomization. Subjects who require or undergo CABG should undergo these procedures a minimum of 4 months in advance of randomization. In addition, subjects who develop a need for revascularization following enrollment should undergo revascularization without delay. Indication for imminent heart transplantation is defined as a high likelihood of transplant prior to collection of the 12 month study endpoint. Candidates cannot be UNOS status 1A or 1B, and they must have documented low probability of being transplanted
2. Valvular heart disease including 1) mechanical or bioprosthetic heart valve; or 2) severe (any valve) insufficiency/regurgitation within 12 months of consent
3. Aortic stenosis with valve area ≤ 1.5 cm2
4. History of ischemic or hemorrhagic stroke within 90 days of consent
5. History of a left ventricular remodeling surgical procedure utilizing prosthetic material
6. Presence of a pacemaker and/or implantable cardioverter-defibrillator (ICD) generator with any of the following limitations/conditions:

   * manufactured before the year 2000
   * leads implanted < 6 weeks prior to consent
   * non-transvenous epicardial, or abandoned leads
   * subcutaneous ICDs
   * leadless pacemakers
   * any other condition that, in the judgment of device-trained staff, would deem an MRI contraindicated
7. Pacemaker-dependence with an ICD (Note: pacemaker-dependent candidates without an ICD are not excluded)
8. A cardiac resynchronization therapy (CRT) device implanted less than 3 months prior to consent
9. Other MRI contraindications (e.g. patient body habitus incompatible with MRI)
10. An appropriate ICD firing or anti-tachycardia pacing (ATP) for ventricular fibrillation or ventricular tachycardia within 30 days of consent
11. Ventricular tachycardia ≥ 20 consecutive beats without an ICD within 3 months of consent, or symptomatic Mobitz II or higher degree atrioventricular block without a functioning pacemaker within 3 months of consent
12. Presence of LV thrombus
13. Evidence of active myocarditis
14. Baseline maximal oxygen consumption (VO2 max) greater than 75% of age and gender based predictive values
15. Baseline eGFR <35 ml/min/1.73m2
16. Blood glucose levels (HbA1c) >10%
17. Hematologic abnormality evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet count < 100,000/ul
18. Liver dysfunction evidenced by enzymes (AST and ALT) ˃ 3 times the upper limit of normal (ULN)
19. Coagulopathy (INR ≥ 1.3) not due to a reversible cause (e.g., warfarin and/or Factor Xa inhibitors). Subjects who cannot be withdrawn from anticoagulation will be excluded.
20. HIV and/or active hepatitis B virus (HBV) or hepatitis C virus (HCV)
21. Allergy to radiographic contrast material that cannot adequately be managed by premedication
22. Known history of anaphylactic reaction to penicillin or streptomycin
23. Received gene or cell-based therapy from any source within the previous 12 months
24. History of malignancy within 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), excluding basal cell carcinoma and cervical carcinoma in situ which have been definitively treated
25. Condition that limits lifespan to < 1 year
26. History of drug abuse (illegal "street" drugs except marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
27. Participation in an investigational therapeutic or device trial within 30 days of consent
28. Cognitive or language barriers that prohibit obtaining informed consent or any study elements
29. Pregnancy or lactation or plans to become pregnant in the next 12 months
30. Any other condition that, in the judgment of the Investigator or Sponsor, would impair enrollment, study product administration, or follow-up

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-10; Primary Completion 2020-06-25 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simari, MD, Study Chair — CCTRN Steering Committee Chair
Locations (7):
- United States (7):
  - Stanford University School of Medicine (Falk Cardiovascular Research Center), Stanford, California
  - University of Florida-Department of Medicine, Gainesville, Florida
  - University of Miami-Interdisciplinary Stem Cell Institute, Miami, Florida
  - Indiana Center for Vascular Biology and Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Hare JM, Bolli R, Cooke JP, Gordon DJ, Henry TD, Perin EC, March KL, Murphy MP, Pepine CJ, Simari RD, Skarlatos SI, Traverse JH, Willerson JT, Szady AD, Taylor DA, Vojvodic RW, Yang PC, Moye LA; Cardiovascular Cell Therapy Research Network. Phase II clinical research design in cardiology: learning the right lessons too well: observations and recommendations from the Cardiovascular Cell Therapy Research Network (CCTRN). Circulation. 2013 Apr 16;127(15):1630-5. doi: 10.1161/CIRCULATIONAHA.112.000779. No abstract available. PMID 23588961
- [Background] Nazarian S, Halperin HR. How to perform magnetic resonance imaging on patients with implantable cardiac arrhythmia devices. Heart Rhythm. 2009 Jan;6(1):138-43. doi: 10.1016/j.hrthm.2008.10.021. Epub 2008 Oct 22. No abstract available. PMID 19121814
- [Background] Bolli R, Hare JM, March KL, Pepine CJ, Willerson JT, Perin EC, Yang PC, Henry TD, Traverse JH, Mitrani RD, Khan A, Hernandez-Schulman I, Taylor DA, DiFede DL, Lima JAC, Chugh A, Loughran J, Vojvodic RW, Sayre SL, Bettencourt J, Cohen M, Moye L, Ebert RF, Simari RD; Cardiovascular Cell Therapy Research Network (CCTRN). Rationale and Design of the CONCERT-HF Trial (Combination of Mesenchymal and c-kit+ Cardiac Stem Cells As Regenerative Therapy for Heart Failure). Circ Res. 2018 Jun 8;122(12):1703-1715. doi: 10.1161/CIRCRESAHA.118.312978. Epub 2018 Apr 27. PMID 29703749
- [Derived] Kato Y, Kizer JR, Ostovaneh MR, Lazar J, Peng Q, van der Geest RJ, Lima JAC, Ambale-Venkatesh B. Extracellular volume-guided late gadolinium enhancement analysis for non-ischemic cardiomyopathy: The Women's Interagency HIV Study. BMC Med Imaging. 2021 Jul 27;21(1):116. doi: 10.1186/s12880-021-00649-6. PMID 34315432
- See also: Cardiovascular Cell Therapy Research Network — http://www.cctrn.org
- See also: National Heart, Lung, and Blood Institute — http://www.nhlbi.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at seven CCTRN centers between November 2016 and November 2018. The main centers are located in Texas, Florida (2 locations), Minnesota, Kentucky, Indiana, and California. Recruitment methods included www.clinicaltrials.gov, local heart failure clinics, and outreach to physician cardiologists. Original sample size of 144 was capped at 125 by NHLBI following review by DSMB of cell production, interim analysis, and power calculations. Power deemed adequate at 125 subjects.
Pre-assignment Details: 125 individuals consented, completed baseline testing, met eligibility criteria, and were randomized to study group. Reasons for failed eligibility (n=68) included investigator discretion, elevated LVEF, MRI contraindications, LV thrombus requiring anticoagulation therapy, elevated peak VO2, and other.
Groups:
- MSCs + CPCs: Target dose of 150 million MSCs and 5 million CPCs
- MSCs: Target dose of 150 million MSCs
- CPCs: Target dose of 5 million CPCs
- Placebo: Plasmalyte A
Period: Overall Study
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Started | 33 | 29 | 31 | 32
Completed | 29 (includes 1 participant who completed final study visit but died within 30 days after final visit.) | 23 | 25 | 25 (includes 1 participant who completed final study visit but died within 30 days after final visit.)
Not Completed | 4 | 6 | 6 | 7
Not completed — Death | 1 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Denominators are of those reporting
Groups:
- Total: Total of all reporting groups
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo | Total
Number analyzed (Participants) | 33 | 29 | 31 | 32 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (11.1) | 61.7 (6.7) | 64.2 (8.1) | 63.1 (8.0) | 62.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 1 | 9
  Male | 31 | 27 | 27 | 31 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 6 | 4 | 20
  Not Hispanic or Latino | 28 | 22 | 25 | 28 | 103
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 2 | 5
  White | 30 | 27 | 28 | 28 | 113
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 31 | 32 | 125
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (3.5) | 30.4 (5.4) | 29.4 (5.0) | 30.0 (4.4) | 30.3 (4.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118.4 (18.2) | 114.0 (11.3) | 117.3 (17.9) | 117.2 (17.6) | 116.8 (16.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 70.2 (9.3) | 70.1 (9.0) | 68.3 (10.8) | 67.7 (11.2) | 69.0 (10.1)
Diabetes [Count of Participants; unit: Participants] — Population: One participant missing data
  Participants
    number analyzed (Participants) | 33 | 28 | 31 | 32 | 124
    (all) | 7 | 10 | 10 | 12 | 39
Hypertension [Count of Participants; unit: Participants] — Population: One participant missing data
  Participants
    number analyzed (Participants) | 33 | 28 | 31 | 32 | 124
    (all) | 29 | 23 | 26 | 27 | 105
Smoking (Lifetime) [Count of Participants; unit: Participants] — Smoking (Lifetime) includes previous and current smokers
  Participants | 19 | 18 | 24 | 22 | 83
Previous Hospitalization for Heart Failure [Count of Participants; unit: Participants] | 11 | 8 | 9 | 13 | 41
Previous Emergency Department Visit for Heart Failure [Count of Participants; unit: Participants] | 6 | 4 | 8 | 9 | 27
Ongoing Ischemia [Count of Participants; unit: Participants] | 9 | 5 | 4 | 7 | 25
New York Heart Association Class 1 [Count of Participants; unit: Participants] — Physician's use the NYHA classification system to place patients into one of four categories based on how much they are limited during physical activity. Class 1 is characterized by no limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 1 | 1 | 3 | 1 | 6
New York Heart Association Class 2 [Count of Participants; unit: Participants] — Physician's use the NYHA classification system to place patients into one of four categories based on how much they are limited during physical activity. Class 2 is characterized by slight limitation of physical activity. The patient is comfortable at rest, however ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 24 | 22 | 26 | 28 | 100
New York Heart Association Class 3 [Count of Participants; unit: Participants] — Physician's use the NYHA classification system to place patients into one of four categories based on how much they are limited during physical activity. Class 3 is characterized by marked limitation of physical activity. The patient is comfortable at rest, however less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Participants | 8 | 6 | 2 | 3 | 19
Presence of a Cardiac Device [Count of Participants; unit: Participants] — Presence of an internal cardiac defibrillator (ICD) or biventricular pacing and ICD.
  Participants | 28 | 24 | 28 | 21 | 101
Number of Myocardial Infarctions [Mean (Standard Deviation); unit: events] — Number of Myocardial Infarctions (lifetime)
  events | 1.6 (1.0) | 1.9 (1.7) | 1.9 (1.2) | 1.7 (1.0) | 1.8 (1.3)
Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] — Variable represents number of patients having undergone PCI procedures (lifetime).
  Participants | 27 | 24 | 27 | 28 | 106
Coronary Artery Bypass Grafting (CABG) [Count of Participants; unit: Participants] — Variable represents the number of patients having undergone a CABG procedure (lifetime).
  Participants | 17 | 14 | 16 | 15 | 62
Multi-Vessel Disease [Count of Participants; unit: Participants] — Multiple vessels supplying blood flow to the left ventricle are affected
  Participants | 25 | 22 | 28 | 30 | 105
Atrial Fibrillation [Count of Participants; unit: Participants] — Variable represents number of patients experiencing atrial fibrillation (lifetime)
  Participants | 11 | 8 | 11 | 10 | 40
Sustained Ventricular Arrhythmia [Count of Participants; unit: Participants] — Variable represents the number of patients experiencing sustained ventricular arrhythmia (lifetime) Population: One participant missing data
  Participants
    number analyzed (Participants) | 32 | 29 | 31 | 32 | 124
    (all) | 12 | 5 | 4 | 7 | 28
Valvular Heart Disease [Count of Participants; unit: Participants] — Variable represents the number of patients diagnosed with valvular heart disease (lifetime)
  Participants | 22 | 17 | 26 | 24 | 89
Beta Blockers [Count of Participants; unit: Participants] — Baseline medications include the use of beta blockers.
  Participants | 32 | 26 | 29 | 31 | 118
ACE Inhibitors [Count of Participants; unit: Participants] — Baseline medications include the use of angiotensin converting enzyme inhibitors (ACE inhibitors)
  Participants | 16 | 10 | 18 | 8 | 52
Angiotensin II Blockers [Count of Participants; unit: Participants] — Baseline medications included the use of angiotensin II blockers
  Participants | 8 | 5 | 6 | 9 | 28
Entresto [Count of Participants; unit: Participants] — Baseline medications included the use of Entresto
  Participants | 8 | 11 | 7 | 13 | 39
Aldosterone Antagonists [Count of Participants; unit: Participants] — Baseline medications included the use of aldosterone antagonists
  Participants | 18 | 20 | 20 | 22 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Change in left ventricular ejection fraction as assessed via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available analyzable LVEF at baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of end diastolic volume
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 28 | 24 | 25 | 25
percentage of end diastolic volume | -0.42 (3.90) | 0.37 (2.95) | 1.05 (3.68) | -0.33 (3.73)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.993, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-2.190 to 2.023], Standard Error of Mean 1.05 — Confidence intervals based on t-test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.499, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-1.229 to 2.635], Standard Error of Mean 0.96 — Confidence intervals based on t-test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.578, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-0.729 to 3.485], Standard Error of Mean 1.05 — Confidence intervals based on t-test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.523, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-3.552 to 0.629], Standard Error of Mean 1.04 — Confidence intervals based on t-test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.471, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-2.7 to 1.127], Standard Error of Mean 0.95 — Confidence intervals based on t-test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.485, ANCOVA; The change in LVEF was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-1.240 to 2.590], Standard Error of Mean 0.95 — Confidence intervals based on t-test

2. Primary Outcome: Change From Baseline in Global Strain (HARP MRI)
Description: Change in global circumferential strain as assessed via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available analyzable global circumferential strain at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 26 | 17 | 22 | 16
percent | -0.36 (3.20) | 0.48 (3.36) | 0.56 (2.08) | -0.10 (3.38)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.942, ANCOVA; The change in global circumferential strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-2.406 to 1.887], Standard Error of Mean 1.05 — Confidence intervals based on t-test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.282, ANCOVA; The change in global circumferential strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-1.815 to 2.975], Standard Error of Mean 1.17 — Confidence intervals based on t-test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.163, ANCOVA; The change in global circumferential strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-1.310 to 2.635], Standard Error of Mean 0.95 — Confidence intervals based on t-test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.175, ANCOVA; The change in global circumferential strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-2.471 to 0.628], Standard Error of Mean 0.77 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.329, ANCOVA; The change in global circumferential strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-2.932 to 1.254], Standard Error of Mean 1.03 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.752, ANCOVA; The change in global circumferential strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-1.829 to 1.994], Standard Error of Mean 0.93 — Confidence intervals based on t-test

3. Primary Outcome: Change From Baseline in Regional Strain (HARP MRI)
Description: Change in regional longitudinal strain as assessed via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available analyzable regional longitudinal strain at baseline and 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 26 | 18 | 22 | 17
percent | -0.50 (2.33) | -0.51 (2.33) | -0.76 (2.49) | -0.91 (2.44)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.733, ANCOVA; The change in regional longitudinal strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-1.118 to 1.927], Standard Error of Mean 0.75 — Confidence intervals based on t-test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.735, ANCOVA; The change in regional longitudinal strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-1.248 to 2.041], Standard Error of Mean 0.81 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.794, ANCOVA; The change in regional longitudinal strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-1.464 to 1.767], Standard Error of Mean 0.80 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.951, ANCOVA; The change in regional longitudinal strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-1.161 to 1.666], Standard Error of Mean 0.70 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.962, ANCOVA; The change in regional longitudinal strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-1.441 to 1.457], Standard Error of Mean 0.71 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.945, ANCOVA; The change in regional longitudinal strain was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.793 to 1.303], Standard Error of Mean 0.76 — Confidence intervals based on t test

4. Primary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVI)
Description: Change in left ventricular end diastolic volume index as measured via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available analyzable LVEDVI at baseline and six months
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 28 | 24 | 25 | 25
mL/m^2 | 0.97 (16.06) | 0.21 (11.91) | -1.13 (12.37) | 2.99 (11.84)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.602, ANCOVA; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -2.02, 95% CI 2-sided [-9.754 to 5.711], Standard Error of Mean 3.85 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.443, ANCOVA; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -2.78, 95% CI 2-sided [-9.609 to 4.044], Standard Error of Mean 3.39 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.348, ANCOVA; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Net) = -4.13, 95% CI 2-sided [-11.011 to 2.760], Standard Error of Mean 3.42 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.812, ANCOVA; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 2.10, 95% CI 2-sided [-5.760 to 9.968], Standard Error of Mean 3.92 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.900, ANCOVA; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-7.052 to 8.574], Standard Error of Mean 3.89 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.848, ANCOVA; The change in LVEDVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-8.321 to 5.635], Standard Error of Mean 3.47 — Confidence intervals based on t test

5. Primary Outcome: Change From Baseline in Left Ventricular End Systolic Volume Index (LVESVI)
Description: Change in left ventricular end systolic volume index as assessed via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available analyzable LVESVI at baseline and 6 months
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 28 | 24 | 25 | 25
mL/m^2 | 0.98 (11.17) | -0.22 (10.75) | -2.37 (11.09) | 2.23 (10.69)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.659, ANCOVA; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-7.281 to 4.789], Standard Error of Mean 3.01 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.466, ANCOVA; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-8.621 to 3.710], Standard Error of Mean 3.06 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.293, ANCOVA; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -4.60, 95% CI 2-sided [-10.799 to 1.594], Standard Error of Mean 3.08 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.530, ANCOVA; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 3.36, 95% CI 2-sided [-2.795 to 9.508], Standard Error of Mean 3.06 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.761, ANCOVA; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-4.910 to 7.330], Standard Error of Mean 3.05 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.669, ANCOVA; The change in LVESVI was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-8.426 to 4.132], Standard Error of Mean 3.12 — Confidence intervals based on t test

6. Primary Outcome: Change From Baseline in Left Ventricular Sphericity Index
Description: Change in left ventricular sphericity as assessed via cardiac MRI. Sphericity index is the ratio of the long and short axis measurements of the left ventricle.
Time Frame: Baseline to 6 months
Population: Participants with available analyzable LV sphericity index at baseline and 6 months
Measure: Mean (Standard Deviation); unit: ratio-unitless
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 26 | 24 | 25 | 25
ratio-unitless | 0.00 (0.07) | -0.00 (0.07) | 0.00 (0.08) | 0.01 (0.08)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.989, ANCOVA; The change in left ventricular sphericity index was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.048 to 0.040], Standard Error of Mean 0.02 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.493, ANCOVA; The change in left ventricular sphericity index was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.056 to 0.033], Standard Error of Mean 0.02 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.926, ANCOVA; The change in left ventricular sphericity index was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.053 to 0.039], Standard Error of Mean 0.02 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.904, ANCOVA; The change in left ventricular sphericity index was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.041 to 0.047], Standard Error of Mean 0.02 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.476, ANCOVA; The change in left ventricular sphericity index was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.035 to 0.049], Standard Error of Mean 0.02 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.515, ANCOVA; The change in left ventricular sphericity index was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.040 to 0.048], Standard Error of Mean 0.02 — Confidence intervals based on t test

7. Primary Outcome: Change From Baseline in Scar Size Percent (DEMRI)
Description: Change in scar size percent as assessed via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available and analyzable scar size data at baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of mass
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 22 | 20 | 22 | 21
percentage of mass | -0.57 (3.25) | -0.70 (2.80) | -1.06 (2.40) | -0.53 (2.29)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.569, ANCOVA; The change in scar size percent was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-1.770 to 1.687], Standard Error of Mean 0.85 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.767, ANCOVA; The change in scar size percent was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-1.792 to 1.457], Standard Error of Mean 0.80 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.261, ANCOVA; The change in scar size percent was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.965 to 0.921], Standard Error of Mean 0.71 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.587, ANCOVA; The change in scar size percent was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-1.261 to 2.222], Standard Error of Mean 0.86 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.994, ANCOVA; The change in scar size percent was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-1.763 to 2.014], Standard Error of Mean 0.93 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.639, ANCOVA; The change in scar size percent was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.993 to 1.283], Standard Error of Mean 0.81 — Confidence intervals based on t test

8. Primary Outcome: Change From Baseline in Scar Tissue Mass (DEMRI)
Description: Change in scar tissue mass as assessed via cardiac MRI
Time Frame: Baseline to 6 months
Population: Participants with available and analyzable scar size data at baseline and 6 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 22 | 20 | 22 | 21
grams | -0.87 (5.21) | -1.13 (3.71) | -2.51 (4.51) | -1.31 (4.07)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.992, ANCOVA; The change in scar tissue mass was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-2.437 to 3.319], Standard Error of Mean 1.42 — Confidence intervals based on t-test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.862, ANCOVA; The change in scar tissue mass was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-2.278 to 2.643], Standard Error of Mean 1.22 — Confidence intervals based on t-test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.217, ANCOVA; The change in scar tissue mass was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-3.846 to 1.443], Standard Error of Mean 1.31 — Confidence intervals based on t-test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.327, ANCOVA; The change in scar tissue mass was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-1.325 to 4.611], Standard Error of Mean 1.47 — Confidence intervals based on t-test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.859, ANCOVA; The change in scar tissue mass was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-2.551 to 3.068], Standard Error of Mean 1.39 — Confidence intervals based on t-test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.338, ANCOVA; The change in scar tissue mass was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-3.952 to 1.184], Standard Error of Mean 1.27 — Confidence intervals based on t-test

9. Primary Outcome: Change From Baseline in Maximal Oxygen Consumption (Peak VO2)
Description: Change in maximal oxygen consumption (peak V02) as assessed via treadmill
Time Frame: Baseline to 6 months
Population: Participants with available analyzable peak VO2 data from baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 28 | 23 | 25 | 26
ml/kg/min | -0.89 (2.94) | -0.83 (3.75) | 0.77 (2.86) | 0.13 (2.28)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.157, ANCOVA; The change in peak VO2 was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-2.456 to 0.411], Standard Error of Mean 0.71 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.428, ANCOVA; The change in peak VO2 was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-2.798 to 0.859], Standard Error of Mean 0.90 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.382, ANCOVA; The change in peak VO2 was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.83 to 2.093], Standard Error of Mean 0.73 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.056, ANCOVA; The change in peak VO2 was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-3.255 to -0.052], Standard Error of Mean 0.80 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.610, ANCOVA; The change in peak VO2 was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-1.991 to 1.885], Standard Error of Mean 0.96 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.195, ANCOVA; The change in peak VO2 was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-0.356 to 3.557], Standard Error of Mean 0.97 — Confidence intervals based on t test

10. Primary Outcome: Change From Baseline in Exercise Tolerance (Six Minute Walk Test)
Description: Change in distance walked (in meters) as measured by the 6 minute walk test. Two walk tests were completed at each endpoint visit (separated by 30 minutes). The average distance of the two walk tests was used for analysis.
Time Frame: Baseline to 6 months
Population: Participants with available analyzable exercise tolerance data at baseline and 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 29 | 24 | 25 | 27
meters | 19.24 (71.65) | 23.85 (57.03) | 2.36 (44.30) | 0.67 (70.54)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.348, ANCOVA; The change in exercise tolerance was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 18.57, 95% CI 2-sided [-19.537 to 56.687], Standard Error of Mean 19.01 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.230, ANCOVA; The change in exercise tolerance was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 23.19, 95% CI 2-sided [-12.759 to 59.134], Standard Error of Mean 17.88 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.905, ANCOVA; The change in exercise tolerance was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [-30.974 to 34.361], Standard Error of Mean 16.21 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.335, ANCOVA; The change in exercise tolerance was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 16.88, 95% CI 2-sided [-15.267 to 49.030], Standard Error of Mean 15.98 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.827, ANCOVA; The change in exercise tolerance was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -4.61, 95% CI 2-sided [-40.106 to 30.880], Standard Error of Mean 17.68 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.163, ANCOVA; The change in exercise tolerance was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -21.49, 95% CI 2-sided [-50.989 to 8.001], Standard Error of Mean 14.63 — Confidence intervals based on t test

11. Primary Outcome: Change From Baseline in Minnesota Living With Heart Failure Questionnaire (MLHFQ) Score
Description: Change in the quality of life summary score as measured by the Minnesota Living with Heart Failure Questionnaire. Minimum and maximum scores for the scale are 0 and 105 respectively. Lower scores indicative of better outcomes.
Time Frame: Baseline to 6 months
Population: Participants with available analyzable MLHFQ summary score at baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 30 | 24 | 25 | 28
score on a scale | -15.32 (16.94) | -20.78 (23.11) | -8.65 (23.72) | -5.68 (18.23)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.023, ANCOVA; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -9.64, 95% CI 2-sided [-18.915 to -0.357], Standard Error of Mean 4.63 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.050, ANCOVA; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -15.09, 95% CI 2-sided [-26.871 to -3.319], Standard Error of Mean 5.84 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.119, ANCOVA; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -2.97, 95% CI 2-sided [-14.784 to 8.836], Standard Error of Mean 5.86 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.845, ANCOVA; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = -6.66, 95% CI 2-sided [-18.087 to 4.762], Standard Error of Mean 5.66 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.976, ANCOVA; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 5.46, 95% CI 2-sided [-5.931 to 16.848], Standard Error of Mean 5.64 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.717, ANCOVA; The change in MLHFQ summary score was compared using ANCOVA analyses adjusting for baseline values; Mean Difference (Final Values) = 12.12, 95% CI 2-sided [-1.337 to 25.578], Standard Error of Mean 6.69 — Confidence intervals based on t test

12. Primary Outcome: Change From Baseline in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP)
Description: Change in N-Terminal pro-Brain Natriuretic Peptide (NT-proBNP) as measured via laboratory blood draw
Time Frame: Baseline to 6 months
Population: Participants with available analyzable NT-proBNP values at baseline and 6 months. Log transformation used. P-values obtained from transformed data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 29 | 23 | 25 | 27
pg/ml | -724.46 (4020.53) | 52.6 (586.16) | 204.09 (533.51) | 687.25 (2006.72)
Statistical Analysis 1: Comparison: MSCs + CPCs vs Placebo; Test type: Superiority; p = 0.110, ANCOVA; Change in NT-proBNP value compared using ANCOVA analyses adjusting for baseline values. Data log transformed, p-values obtained from transformed data; Mean Difference (Final Values) = -1411.7, 95% CI 2-sided [-3108.3 to 284.9], Standard Error of Mean 840.6 — Confidence intervals based on t test
Statistical Analysis 2: Comparison: MSCs vs Placebo; Test type: Superiority; p = 0.112, ANCOVA; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -634.6, 95% CI 2-sided [-1460.7 to 191.4], Standard Error of Mean 405.1 — Confidence intervals based on t test
Statistical Analysis 3: Comparison: CPCs vs Placebo; Test type: Superiority; p = 0.891, ANCOVA; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -483.2, 95% CI 2-sided [-1301.5 to 335.2], Standard Error of Mean 400.7 — Confidence intervals based on t test
Statistical Analysis 4: Comparison: MSCs + CPCs vs CPCs; Test type: Superiority; p = 0.009, ANCOVA; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -928.6, 95% CI 2-sided [-2470.7 to 613.6], Standard Error of Mean 754.2 — Confidence intervals based on t test
Statistical Analysis 5: Comparison: MSCs + CPCs vs MSCs; Test type: Superiority; p = 0.661, ANCOVA; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -777.1, 95% CI 2-sided [-2323.2 to 769.1], Standard Error of Mean 756.5 — Confidence intervals based on t test
Statistical Analysis 6: Comparison: MSCs vs CPCs; Test type: Superiority; p = 0.015, ANCOVA; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = 151.5, 95% CI 2-sided [-175.4 to 478.4], Standard Error of Mean 162.2 — Confidence intervals based on t test

13. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)-Trajectory
Description: The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). The first set of results reflects the model within each arm and represents change per 6 months within that treatment arm. The second set of results reflects an overall model with all patients and the results represent the change per 6 months irrespective of treatment arm.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable LVEF at baseline, 6 months, and 12 months.
Measure: Least Squares Mean (Standard Error); unit: percentage of end diastolic volume
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
percentage of end diastolic volume | 0.167 (0.551) | 0.422 (0.480) | 0.633 (0.411) | -0.175 (0.332)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; Repeated-measures linear regression models were used to address trajectories (upward or downward trends) over time within each of the 4 treatment groups. Results of the overall model are reported; Test type: Other; p = 0.269, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 0.267, Standard Error of Mean 0.241 — "Standard error of the mean" is the standard error of the estimate of the slope of time

14. Primary Outcome: Change From Baseline in Global Strain (HARP MRI)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had available analyzable global circumferential strain at baseline, 6 month, and 12 month.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
percent | 0.126 (0.239) | -0.324 (0.283) | 0.276 (0.300) | 0.576 (0.417)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.361, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 0.141, Standard Error of Mean 0.153 — "Standard error of the mean" is the standard error of the estimate of the slope of time

15. Primary Outcome: Change From Baseline in Regional Strain (HARP MRI)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable regional strain at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
percent | -0.084 (0.287) | -0.385 (0.350) | -0.325 (0.323) | -0.288 (0.360)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.107, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = -0.267, Standard Error of Mean 0.164 — "Standard error of the mean" is the standard error of the estimate of the slope of time

16. Primary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVI)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable LVEDVI at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: mL/m^2
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
mL/m^2 | 1.538 (1.585) | 0.320 (1.303) | 1.796 (1.393) | 1.862 (1.980)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.095, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 1.395, Standard Error of Mean 0.829 — "Standard error of the mean" is the standard error of the estimate of the slope of time

17. Primary Outcome: Change From Baseline in Left Ventricular End Systolic Volume Index (LVESVI)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, 12 months)
Population: Participants who had analyzable LVESVI at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: mL/m^2
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
mL/m^2 | 0.826 (1.158) | -0.394 (1.117) | 0.626 (1.288) | 1.077 (1.709)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.379, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 0.603, Standard Error of Mean 0.683 — "Standard error of the mean" is the standard error of the estimate of the slope of time

18. Primary Outcome: Change From Baseline in Left Ventricular Sphericity Index-Trajectory
Description: Sphericity index is the ratio of the long and short axis measurements of the left ventricle. The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). The first set of results reflects the model within each arm and represents change per 6 months within that treatment arm. The second set of results reflects an overall model with all patients and the results represent the change per 6 months irrespective of treatment arm.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable LV Sphericity Index at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: ratio-unitless
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
ratio-unitless | 0.004 (0.007) | -0.004 (0.008) | 0.008 (0.007) | 0.002 (0.012)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.401, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 0.003, Standard Error of Mean 0.004 — "Standard error of the mean" is the standard error of the estimate of the slope of time

19. Primary Outcome: Change From Baseline in Scar Size Percent (DEMRI)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable scar size percent at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: percentage of mass
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
percentage of mass | -0.341 (0.314) | -0.290 (0.231) | -0.427 (0.306) | -0.013 (0.340)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.126, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = -0.244, Standard Error of Mean 0.158 — "Standard error of the mean" is the standard error of the estimate of the slope of time

20. Primary Outcome: Change From Baseline in Scar Tissue Mass (DEMRI)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable scar size data at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
grams | -0.309 (0.539) | -0.266 (0.367) | -0.958 (0.615) | -0.390 (0.549)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.139, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = -0.420, Standard Error of Mean 0.281 — "Standard error of the mean" is the standard error of the estimate of the slope of time

21. Primary Outcome: Change From Baseline in Maximal Oxygen Consumption (Peak VO2)-Trajectory
Description: as for outcome 13
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable peak VO2 at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: ml/kg/min
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
ml/kg/min | -0.711 (0.352) | 0.632 (0.275) | -0.165 (0.325) | -0.093 (0.369)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.472, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = -0.133, Standard Error of Mean 0.184 — "Standard error of the mean" is the standard error of the estimate of the slope of time

22. Primary Outcome: Change From Baseline in Exercise Tolerance (Six Minute Walk Test)-Trajectory
Description: Two walk tests were completed at each endpoint visit (separated by 30 minutes). The average distance of the two walk tests was used for analysis. The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). The first set of results reflects the model within each arm and represents change per 6 months within that treatment arm. The second set of results reflects an overall model with all patients and the results represent the change per 6 months irrespective of treatment arm.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable six minute walk tests at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
meters | 9.996 (5.558) | 11.434 (5.531) | 6.776 (6.192) | -4.248 (5.215)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.025, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 6.544, Standard Error of Mean 2.882 — "Standard error of the mean" is the standard error of the estimate of the slope of time

23. Primary Outcome: Change From Baseline in Minnesota Living With Heart Failure Questionnaire (MLHFQ) Score-Trajectory
Description: Minimum and maximum scores for the scale are 0 and 105 respectively. Lower scores indicative of better outcomes. The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). The first set of results reflects the model within each arm and represents change per 6 months within that treatment arm. The 2nd and 3rd set of results represent differences for varying slopes from the interaction model.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable MLHFQ scores at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
score on a scale | -9.258 (2.079) | -7.295 (2.746) | 0.776 (1.731) | -2.378 (2.357)
Statistical Analysis 1: Comparison: MSCs vs Placebo; Repeated-measures linear regression models were used to address trajectories (upward or downward trends) over time within each of the 4 treatment groups. A time by treatment interaction was assessed; Test type: Other; p = 0.037, Regression, Linear; slope with interaction = -7.08, Standard Error of Mean 3.3
Statistical Analysis 2: Comparison: MSCs + CPCs vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Other; p = 0.035, Regression, Linear; slope with interaction = -6.78, Standard Error of Mean 3.18

24. Primary Outcome: Change From Baseline in N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP)-Trajectory
Description: Log transformation used. The change in this measure over time is assessed using a repeated measures linear regression model of trajectory (change over time). The first set of results reflects the model within each arm and represents change per 6 months within that treatment arm. The second set of results reflects an overall model with all patients and the results represent the change per 6 months irrespective of treatment arm.
Time Frame: Assessed as a trajectory (baseline, 6 months, and 12 months)
Population: Participants who had analyzable NT-proBNP values at baseline, 6 months, and 12 months
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
pg/ml | 74.650 (72.303) | 102.250 (46.194) | 61.680 (57.365) | 185.210 (99.190)
Statistical Analysis 1: Comparison: MSCs + CPCs vs MSCs vs CPCs vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.092, Repeated Measures Linear Regression — No adjustments for multiplicity were made in this Phase II trial; slope of time = 84.557, Standard Error of Mean 35.810 — "Standard error of the mean" is the standard error of the estimate of the slope of time

25. Primary Outcome: Participants With Major Adverse Cardiac Events (MACE)
Description: Number of participants with adjudicated events including death, hospitalization for worsening heart failure, and/or other exacerbation of heart failure (non-hospitalization).
Time Frame: Baseline to End of 12 Month Visit Window, an average of 395 days following study product injection
Population: Population includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
Participants | 3 | 7 | 2 | 9

26. Primary Outcome: Participants Experiencing Other Significant Clinical Events
Description: Number of participants experiencing other significant adjudicated clinical events including: non-fatal stroke, non-fatal MI, coronary artery revascularization, ventricular tachycardia/fibrillation, and pericardial tamponade
Time Frame: Baseline to End of 12 Month Visit Window, an average of 395 days following study product injection
Population: Population includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
Participants | 8 | 3 | 11 | 7

27. Primary Outcome: Cumulative Days Alive and Out of Hospital for Heart Failure
Description: Days alive and out of hospital during the study evaluation period. Subjects were allotted a visit window extending 30 days past their anticipated 12-month visit. Some participants had extended 12-month visit windows due to the COVID-19 pandemic.
Time Frame: Baseline to End of 12 Month Visit Window, an average of 395 days following study product injection
Population: Comparison of the 4 treatment groups on days alive and out of the hospital for heart failure during the 12 month study evaluation period; adjusted for time in followup. Analysis includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
days | 472 (121) | 448 (120) | 438 (163) | 427 (158)

28. Other Pre Specified Outcome: Subjects With Events Between Randomization and Study Product Injection (SPI) That Preclude the Receipt of Product
Description: Number and percent of subjects with events between randomization and study product injection (SPI) that preclude the subject from receiving product. Reasons include those who did not undergo harvest (n=6; death, subject withdraw, subject changed mind) and those who did not undergo SPI (n=9; death, LVAD placement, episodes of ventricular tachycardia, and cancelled procedures)
Time Frame: Randomization to SPI, an average of 14 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 29 | 31 | 32
Participants | 3 | 4 | 4 | 4

29. Other Pre Specified Outcome: Subjects Who Have a Failed Bone Marrow Aspiration Procedure
Description: Number and percent of subjects who do not successfully undergo bone marrow aspiration
Time Frame: During bone marrow aspiration procedure
Population: Participants who attended their harvest visit
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 27 | 30 | 29
Participants | 0 | 0 | 0 | 0

30. Other Pre Specified Outcome: Subjects Who Have a Failed Endomyocardial Biopsy Procedure
Description: Number and percent of subjects who do not successfully undergo endomyocardial biopsy procedure. Note only participants who were assigned to MSC+CPC or to CPC groups had endomyocardial biopsy procedures attempted.
Time Frame: During endomyocardial biopsy procedure
Population: Participants who attended the harvest visit and were assigned to either MSCs+CPCs or CPCs.
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 33 | 0 | 30 | 0
Participants | 0 | 0 | 1 | 0

31. Other Pre Specified Outcome: Subject MSC Products Which Failed Release Criteria
Description: Number and percent of subjects who have MSC products which failed release criteria
Time Frame: Harvest to Study Product Injection Procedure
Population: Population includes only those participant products assigned to treatment groups including MSCs.
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 30 | 25 | 0 | 0
Participants | 8 | 6 |  |

32. Other Pre Specified Outcome: Subject CPC Products Which Failed Release Criteria
Description: Number and percent of subjects who have CPC products which failed release criteria
Time Frame: Harvest to Study Project Injection procedure
Population: Population includes only those participant products assigned to treatment groups including CPCs.
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 30 | 0 | 27 | 0
Participants | 5 |  | 4 |

33. Other Pre Specified Outcome: Subjects Who Receive Less Than 15 Injections During SPI
Description: Number and percent of subjects who received less than 15 injections during SPI
Time Frame: During SPI procedure
Population: Participants who received study product administration
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 30 | 25 | 27 | 28
Participants | 2 | 0 | 1 | 1

34. Other Pre Specified Outcome: Subjects Who Have at Least One Cardiac MRI Endpoint Measure That is Uninterpretable
Description: Number and percent of subjects who have at least one cardiac MRI endpoint measure that is uninterpretable due to issues related to the device, including, but not limited to, inability to undergo the procedure
Time Frame: Baseline to 12 months
Population: Participants completing an MRI scan at both baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
Number analyzed (Participants) | 29 | 20 | 23 | 22
Participants | 5 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: Events reported occurred between randomization and the end of 12 Month Visit Window (an average of 395 days following study product injection).
Description: Events were assessed systematically at each study visit during the physical exam assessment. A standard workbook was used to collect event details. Sponsor safety team reviewed events and requested additional documentation as needed.
Arm/Group | MSCs + CPCs | MSCs | CPCs | Placebo
All-Cause Mortality (participants affected / at risk) | 2/33 | 3/29 | 2/31 | 4/32
Serious Adverse Events (participants affected / at risk) | 14/33 | 14/29 | 13/31 | 18/32
Other Adverse Events (participants affected / at risk) | 10/33 | 6/29 | 14/31 | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSCs + CPCs (N=33) | MSCs (N=29) | CPCs (N=31) | Placebo (N=32)
Anaemia or Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Angina pectoris or angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 3 (4) | 3 (4) | 1 (2) | 10 (20)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 5 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device lead damage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular assist device insertion (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSCs + CPCs (N=33) | MSCs (N=29) | CPCs (N=31) | Placebo (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Angina pectoris or angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 5 (6) | 0 (0) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Relatively small group sizes overall. Relatively long interval between harvest visit and study product injection (approx. 14wks) resulting in patient attrition. Failure of cells to grow from tissue of some patients, resulting in some patients crossing over into other treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02501811/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT02501811/Prot_SAP_001.pdf